CLINICAL TRIAL: NCT06350799
Title: COPD Home-Visits: Community Health Worker Home-visit Support to Enhance Self-Management and Improve Quality of Life Among Rural Veterans With Chronic Obstructive Pulmonary Disease
Brief Title: Chronic Obstructive Pulmonary Disease and Community Health Worker Home-visits
Status: Completed | Type: Observational
Sponsor: VA Puget Sound Health Care System (U.S. Federal Agency)
Collaborators: Public Health - Seattle and King County (Other Government); University of Washington (Other)
Responsible Party: Principal Investigator, Vincent S. Fan, Principal Investigator, VA Puget Sound Health Care System
Other Study IDs: 01741
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: COPD
Keywords: Community Health Workers
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We examined a Community Health Worker (CHW) program for Chronic Obstructive Pulmonary Disease (COPD) in Veteran Participants. The goal of this study was to assess participants' perceived acceptability, appropriateness, and feasibility of the intervention, explore participants' COPD health outcomes, and gather insights from participants and CHWs to inform potential improvements.

Veteran participants enrolled in the 12-week intervention and received a series of 9 CHW home, phone, or video visits. These visits provided education and chronic disease self-management practices to improve COPD health.

Researchers examined the participant and CHW perception of the intervention through qualitative interviews and surveys.

DETAILED DESCRIPTION:
Background: One-third of Veterans live in rural areas, and rural patients are more likely to have chronic obstructive pulmonary disease (COPD) and rural Veterans with COPD have lower health status than urban Veterans. COPD patients often have exacerbations that can lead to emergency room visits and hospitalizations. Since COPD exacerbations and hospitalizations can be prevented by interventions such as appropriate use of inhaled COPD medications, focusing efforts to improve COPD management for these high-risk rural Veterans with COPD is essential.

Objectives: The proposed project will test the feasibility and potential effectiveness of a Community Health Worker (CHW) intervention to help reduce risk of COPD exacerbations among Veterans. The overall goal of this pilot study is to determine the feasibility and acceptability of a community health worker intervention to promote health behavior change among Veterans with COPD. To target a high risk population, we will focus on Veterans with moderate-severe exacerbations in the past year.

Methods: Participants at VA Puget Sound will be enrolled in the study. We will develop a program to serve rural Veterans, though we will also serve all Veterans meeting the criteria particularly in these initial stages at the VA Puget Sound in Seattle. Participants will be scheduled for 9 education visits over 12 weeks that will be delivered either in-person, though a Clinical Video Telehealth into the home (CVT-to-Home), or by phone. Participants will be offered to have additional phone calls in between visits to check-in on their COPD self-management goals and confirm their upcoming appointments. Participants will be followed for a total of 3 months in this pilot study. Data on proportion of eligible patients who enroll in the study, number of intervention visits completed, and completion of study questionnaires will be collected. Data analysis will examine whether any changes in outcomes such as quality of life or physical activity between baseline and follow-up are associated with the intervention. Semi-structured exit interviews will be conducted at the end of the study to assess the design of intervention components, use of technology, appropriateness, and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of COPD
* Enrolled in VA primary care
* English speaking
* Access to a telephone
* Clinically stable breathing for at least 1 month prior to enrollment
* If available, post-bronchodilator spirometry with FEV1/FVC < 0.70 in the last 5 years
* ≥ 1 exacerbation in the past year treated with prednisone and/or antibiotics or treated in the ED or stay in the hospital
* Ability to connect to CVT-to-Home

Exclusion Criteria:

* Nursing home resident or institutionalized
* Pregnancy
* Pulmonary rehabilitation program in the last year
* Uncontrolled hypertension, angina, or heart failure
* Life expectancy < 1 year or terminal illness.
* Dementia or uncontrolled psychiatric illness
* Other safety concerns with participating in physical activity

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients recruited for this study will be Veterans with COPD.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2019-03-14 (Actual); Primary Completion 2021-05-27 (Actual); Study Completion 2023-04-28 (Actual)

PRIMARY OUTCOMES:
Acceptability, Appropriateness, Feasibility | one month post-intervention
  Patient perception through interviews

CONTACTS AND LOCATIONS:
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No